CLINICAL TRIAL: NCT06515834
Title: A Placebo-controlled, Within-group Randomised, and Double-blind Trial Investigating Safety, Tolerability, and Pharmacokinetics of FE 999301 After Single Ascending Doses in Healthy Japanese Men
Brief Title: Investigating the Safety, Tolerability, Immunogenicity and Pharmacokinetics of Olamkicept in Healthy Japanese Persons
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 000435
Record Dates: First submitted 2024-07-01; First posted 2024-07-23 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-07

CONDITIONS: Gastroenterology

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- FE 999301 (Active Comparator)
  Interventions: Drug: FE 999301

INTERVENTIONS:
Drug: FE 999301 — To assess the safety and tolerability of FE 999301 after single intravenous (IV) dose infusion in healthy Japanese men
  Arms: FE 999301
Drug: Placebo — Placebo to assess the safety and tolerability of FE 999301 after single intravenous (IV) dose infusion in healthy Japanese men
  Arms: Placebo

SUMMARY:
Interleukin (IL)-6 is a cytokine produced in response to infection and tissue damage. IL-6 is believed to act as a key mediator in chronic inflammation and autoimmune diseases such as inflammatory bowel diseases. IL-6 is known to be involved in at least two distinct signalling pathways, classical and trans-signalling. The hypothesis is that classical signalling by IL-6 infers some beneficial effects (e.g. on gut barrier function), while excessive IL-6 trans-signalling may have detrimental effects. Olamkicept (FE 999301) has been shown in vitro to be a selective IL-6 trans-signalling inhibitor and administered at lower doses, it has proven to induce clinical improvement for patients with ulcerative colitis. The aim of this trial is to investigate safety, tolerability, immunogenicity and pharmacokinetics of Olamkicept at higher doses, to support the clinical development program. The hypothesis for this study is that treatment with higher doses of Olamkicept will result in greater clinical improvement for participants with inflammatory bowel diseases.

ELIGIBILITY:
Inclusion Criteria:

* In good health, determined by:

  * no clinically significant findings from medical history,
  * physical examination,
  * 12-lead electrocardiogram (ECG),
  * vital signs measurements,
  * and clinical laboratory evaluations

Exclusion Criteria:

* History of clinically significant medical conditions including, but not limited to:

  * diseases of the renal,
  * hepatic,
  * respiratory,
  * gastrointestinal,
  * cardiovascular,
  * neurological,
  * musculoskeletal,
  * immunological,
  * haematological,
  * endocrine,
  * and metabolic systems,
  * as well as oncological,
  * psychiatric,
  * dermatological,
  * and allergic diseases (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Number treatment-emergent adverse events | From baseline up to 36 days after a single dose infusion
  Number of treatment-emergent adverse events, including type, intensity, and causality
Blood pressure | From baseline up to 36 days after a single dose infusion
  Change from baseline in vital signs comprising systolic and diastolic blood pressure
Pulse | From baseline up to 36 days after a single dose infusion
  Change from baseline in vital signs comprising pulse
Body temperature | From baseline up to 36 days after a single dose infusion
  Change from baseline in vital signs comprising body temperature
Heart rate | From baseline up to 36 days after a single dose infusion
  Change from baseline in 12-lead electrocardiogram (ECG) assessing heart rate after a single IV dose infusion.
PR interval | From baseline up to 36 days after a single dose infusion
  Change from baseline in 12-lead electrocardiogram ECG assessing the PR interval after a single IV dose infusion.
RR interval | From baseline up to 36 days after a single dose infusion
  Change from baseline in 12-lead ECG assessing the RR interval after a single IV dose infusion.
QRS duration | From baseline up to 36 days after a single dose infusion
  Change from baseline in 12-lead ECG assessing QRS duration after a single IV dose infusion.
QT interval | From baseline up to 36 days after a single dose infusion
  Change from baseline in 12-lead ECG assessing QT interval after a single IV dose infusion.
QTc interval | From baseline up to 36 days after a single dose infusion
  Change from baseline in 12-lead electrocardiogram (ECG) assessing QTc interval after a single IV dose infusion.
QRS axis | From baseline up to 36 days after a single dose infusion
  Change from baseline in 12-lead ECG assessing QRS axis after a single IV dose infusion.
Change in haematology | From baseline up to 36 days after a single dose infusion
  Number of participants with clinically significant abnormal findings in haematology (haematocrit, haemoglobin, mean cellular volume (MCV), mean corpuscular haemoglobin content (MCHC), platelet count, red blood cell count, reticulocytes, white blood cell count with differential count, neutrophils, eosinophils, basophils, lymphocytes, monocytes) from baseline up to and including Day 36 after a single dose infusion.
Clinical chemistry | From baseline up to 36 days after a single dose infusion
  Number of participants with clinically significant abnormal findings in clinical chemistry (alanine aminotranferase (ALT), albumin, alkaline phosphatase, aspartate aminotranferase (AST), glucose, calcium, chloride, cholesterol, C-reactive protein, creatinine, estimated glomerular filtration rate (eGFR), gamma-glutamyltranferase, phosphate, potassium, sodium, thyroid stimulating hormone, free triiodothyronine, free thyroxine, total bilirubin, urea (blood urea nitrogen)), from baseline up to and including Day 36 after a single dose infusion.
Haemostasis | From baseline up to 36 days after a single dose infusion
  Blood and urine samples to assess change from baseline in haemostasis after a single IV dose infusion.
Protein urinalysis parameter | From baseline up to 36 days after a single dose infusion
  Number of participants with clinically significant abnormal findings in protein urinalysis parameter from baseline up to and including Day 36 after a single dose infusion.
Glucose urinalysis parameter | From baseline up to 36 days after a single dose infusion
  Number of participants with clinically significant abnormal findings in glucose urinalysis parameter from baseline up to and including Day 36 after a single dose infusion.
Bilirubin urinalysis parameter | From baseline up to 36 days after a single dose infusion
  Number of participants with clinically significant abnormal findings in bilirubin urinalysis parameter from baseline up to and including Day 36 after a single dose infusion.
pH urinalysis parameter | From baseline up to 36 days after a single dose infusion
  Number of participants with clinically significant abnormal findings in pH urinalysis parameter from baseline up to and including Day 36 after a single dose infusion.
Nitrate urinalysis parameter | From baseline up to 36 days after a single dose infusion
  Number of participants with clinically significant abnormal findings in nitrate urinalysis parameter from baseline up to and including Day 36 after a single dose infusion.
Ketone urinalysis parameter | From baseline up to 36 days after a single dose infusion
  Number of participants with clinically significant abnormal findings in ketone urinalysis parameter from baseline up to and including Day 36 after a single dose infusion.
Urobilinogen urinalysis parameter | From baseline up to 36 days after a single dose infusion
  Number of participants with clinically significant abnormal findings in urobilinogen urinalysis parameter from baseline up to and including Day 36 after a single dose infusion.
Blood urinalysis parameter | From baseline up to 36 days after a single dose infusion
  Number of participants with clinically significant abnormal findings in blood urinalysis parameter from baseline up to and including Day 36 after a single dose infusion.
Leukocyte urinalysis parameter | From baseline up to 36 days after a single dose infusion
  Number of participants with clinically significant abnormal findings in leukocyte urinalysis parameter from baseline up to and including Day 36 after a single dose infusion.
Specific gravity urinalysis parameter | From baseline up to 36 days after a single dose infusion
  Number of participants with clinically significant abnormal findings in specific gravity urinalysis parameter from baseline up to and including Day 36 after a single dose infusion.

SECONDARY OUTCOMES:
Area under the Curve to Infinity (AUCinf) | From baseline up to 36 days after a single dose infusion
  Single-dose Pharmacokinetics of FE 999301 evaluating the AUCinf after single IV dose infusion in healthy Japanese men.
Area Under the Curve last concentration (AUClast) | From baseline up to 36 days after a single dose infusion
  Single-dose Pharmacokinetics of FE 999301 evaluating AUClast after single IV dose infusion in healthy Japanese men.
Concentration at the end of infusion (Ceoi) | From baseline up to 36 days after a single dose infusion
  Single-dose Pharmacokinetics of FE 999301 assessing Ceoi after single IV dose infusion in healthy Japanese men.
Maximum concentration (Cmax) | From baseline up to 36 days after a single dose infusion
  Single-dose Pharmacokinetics of FE 999301 evaluating maximum concentration in the body Cmax after a single IV dose infusion in healthy Japanese men.
Time to reach maximum concentration (tmax) | From baseline up to 36 days after a single dose infusion
  Single-dose Pharmacokinetics of FE 999301 evaluating time to reach the maximum concentration in the body after a single IV dose infusion in healthy Japanese men.
Elimination half-life (t1/2) | From baseline up to 36 days after a single dose infusion
  Single-dose Pharmacokinetics of FE 999301 evaluating the amount of time required for the drug concentration to be reduced to exactly half of its initial concentration in the blood after single IV dose infusion in healthy Japanese men.
Mean residence time (MRT) | From baseline up to 36 days after a single dose infusion
  Single-dose Pharmacokinetics of FE 999301 assessing the average time the drug stays in the body after single IV dose infusion in healthy Japanese men.
Clearance (CL) | From baseline up to 36 days after a single dose infusion
  Single-dose Pharmacokinetics of FE 999301 evaluating the rate at which the drug is removed from the body after single IV dose infusion in healthy Japanese men.
Volume of Distribution at steady state (Vss) | From baseline up to 36 days after a single dose infusion
  Single-dose Pharmacokinetics of FE 999301 assessing the volume of distribution at a steady state after single IV dose infusion in healthy Japanese men.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Ferring Investigational Site, Sumida-Ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No